CLINICAL TRIAL: NCT04735887
Title: The Impact of an Evidence-Informed Spinal Cord Injury Activities of Daily Living Educational Manual (SADL-eM): Study Protocol for a Randomized Clinical Trial
Brief Title: The Impact of an Evidence-Informed Spinal Cord Injury Activities of Daily Living Educational Manual
Acronym: SADLeM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Moussa Abu Mostafa, Principal investigator, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 972225221
Record Dates: First submitted 2021-01-22; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injuries
Keywords: Occupational therapy; educational intervention; Activities of daily living; Spinal Cord Injury; clinical trials
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The research assistant who will perform data collection will be blinded to the patient group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SADL-eM & conventional therapy (Experimental): Patients with SCI treated in an inpatient rehabilitation setting who receive a copy of the SADL-eM in addition to conventional therapy.
  Interventions: Other: SADL-eM
- Conventional therapy (No Intervention): Patients with SCI treated in an inpatient rehabilitation setting who receive conventional therapy.

INTERVENTIONS:
Other: SADL-eM — The SADL-eM includes three elements essential to the intervention, namely: knowledge, skills, and advice. The manual includes 92 A5 pages with six detailed sections: an Introduction and five chapters: (1) Rehabilitation team, (2) Activities of Daily Living, (3) Assistive devices, (4) Home environment adaptation, and (5) Knowledge guide. The SADL-eM uses text and illustrative pictures that are carefully selected for contextual relevance. The manual is simple, easy, and suitable for people with a non-medical background.
  Other Names: Spinal Cord Injury Activities of Daily Living Educational Manual
  Arms: SADL-eM & conventional therapy

SUMMARY:
This study argues that providing evidence-based occupational therapy patient education is vital in order to optimize rehabilitation outcomes. The planned trial aims to evaluate the SADL-eM intervention for people with SCI compared with standard treatment.

DETAILED DESCRIPTION:
This is a parallel randomized clinical trial with two study arms, intervention and control. Ninety patients treated in three inpatient rehabilitation settings will be randomly allocated to two study groups. Both groups will receive standard care. The intervention group will also receive a copy of the SADL-eM from their treating occupational therapist during an individual session. Assessment on admission (baseline measure) and after six weeks of admission will use the SCIM-SR as the primary outcome measure. Secondary outcomes include the SCIM-III, Private Religiousness Practices Scale, Organizational Religiousness Short-Form, additional domains of ADL covered by the educational manual, and adherence to the intervention. The effect will be determined using repeated-measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SCI diagnosis by computed tomography or magnetic resonance report.
* ASIA: A, B, and C
* Age between 18 and 65 years old.
* Stable medical condition.
* Time elapsed after SCI is not more than 6 months.
* Minimum time of stay in the inpatient rehabilitation unit is six weeks.
* Active involvement in the rehabilitation program.
* Sufficient comprehension (read/write) of the Arabic language.

Exclusion Criteria:

* Unconfirmed diagnosis.
* Patients who have communication and/or cognitive disorders such as global aphasia and memory deficit.
* Patients with a disturbed level of awareness such as coma or lethargy.
* Time elapsed since SCI is more than 6 months.
* ASIA: D and E
* Unstable medical condition.
* Patients who have other cause(s) of disability in addition to SCI such as stroke or amputation.
* Age less than 18 or more than 65 years old.
* Time of stay in the inpatient rehabilitation unit is less than six weeks.
* Inactive involvement in the rehabilitation program.
* Patients with progressive disease or a psychiatric condition that would interfere with active participation in the rehabilitation programs.
* Patients with cardiovascular contraindications.
* Persons who become walking ambulatory during the inpatient period.
* Persons with complete tetraplegia C4 or above.
* Persons on a mechanical ventilator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Independence Measure-Self Reported (SCIM-SR) baseline assessment | within 3 days of admission
  Spinal Cord Independence Measure-Self Reported is a patient-reported 17-item tool that evaluates the ability of a person with SCI to perform specified activities independently, with assistance, or with assistive devices. Total score ranges between 0-100, higher scores mean better.
Spinal Cord Independence Measure-Self Reported (SCIM-SR) change after six weeks | Six weeks after admission
  Spinal Cord Independence Measure-Self Reported is a patient-reported 17-item tool that evaluates the ability of a person with SCI to perform specified activities independently, with assistance, or with assistive devices. Total score ranges between 0-100, higher scores mean better.

SECONDARY OUTCOMES:
Spinal Cord Independence Measure-III (SCIM-III) baseline assessment | within 3 days of admission
  Spinal Cord Independence Measure-III is a 17-task tool that evaluates the ability of a person with SCI to perform specified activities independently, with assistance, or with assistive devices. It is therapist-reported. Total score ranges between 0-100, higher scores mean better.
Spinal Cord Independence Measure-III (SCIM-III) change after six weeks | Six weeks after admission
  Spinal Cord Independence Measure-III is a 17-task tool that evaluates the ability of a person with SCI to perform specified activities independently, with assistance, or with assistive devices. It is therapist-reported. Total score ranges between 0-100, higher scores mean better.

CONTACTS AND LOCATIONS:
Overall Officials: Moussa Abu Mostafa, Master, Principal Investigator — Hamad Rehabilitation Hospital
Locations (3):
- Palestinian Territories (3):
  - Hamad Rehabilitation Hospital, Gaza, Gaza Strip
  - ElAmal Rehabilitation Hospital, Khan Yunis, Gaza Strip
  - ElWafa Rehabilitation Hospital, Zahra City, Gaza Strip

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available. Data collected will be used only for analysis and results production.

REFERENCES:
- [Background] Magill N, Knight R, McCrone P, Ismail K, Landau S. A scoping review of the problems and solutions associated with contamination in trials of complex interventions in mental health. BMC Med Res Methodol. 2019 Jan 7;19(1):4. doi: 10.1186/s12874-018-0646-z. PMID 30616508
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Bodling, A., Heneghan, M., Walsh, J. C., Yoon, D. P., & Johnstone, B. (2013). The brief multidimensional measure of religiousness/spirituality with an irish sample: A factor analysis. International Journal of Therapy and Rehabilitation, 20(2), 72-78. https://doi.org/10.12968/ijtr.2013.20.2.72
- [Background] De Las Cuevas C, Penate W. Psychometric properties of the eight-item Morisky Medication Adherence Scale (MMAS-8) in a psychiatric outpatient setting. Int J Clin Health Psychol. 2015 May-Aug;15(2):121-129. doi: 10.1016/j.ijchp.2014.11.003. Epub 2014 Dec 25. PMID 30487829
- [Background] DiSilvio B, Virani A, Patel S, Finoli L, Singh A, DuMont T, Cheema T. Institutional COVID-19 Protocols: Focused on Preparation, Safety, and Care Consolidation. Crit Care Nurs Q. 2020 Oct/Dec;43(4):413-427. doi: 10.1097/CNQ.0000000000000327. PMID 32833778
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fekete C, Eriks-Hoogland I, Baumberger M, Catz A, Itzkovich M, Luthi H, Post MW, von Elm E, Wyss A, Brinkhof MW. Development and validation of a self-report version of the Spinal Cord Independence Measure (SCIM III). Spinal Cord. 2013 Jan;51(1):40-7. doi: 10.1038/sc.2012.87. Epub 2012 Aug 14. PMID 22890418
- [Background] Krueger C, Tian L. A comparison of the general linear mixed model and repeated measures ANOVA using a dataset with multiple missing data points. Biol Res Nurs. 2004 Oct;6(2):151-7. doi: 10.1177/1099800404267682. PMID 15388912
- [Background] Fetzer Institute, N. I. on A. W. G. (2003). Multidimensional Measurement of Religiousness/ Spirituality for Use in Health Research: A Report of the Fetzer Institute/ National Institute on Aging Working Group.
- [Background] Glass CA, Tesio L, Itzkovich M, Soni BM, Silva P, Mecci M, Chadwick R, el Masry W, Osman A, Savic G, Gardner B, Bergstrom E, Catz A. Spinal Cord Independence Measure, version III: applicability to the UK spinal cord injured population. J Rehabil Med. 2009 Sep;41(9):723-8. doi: 10.2340/16501977-0398. PMID 19774305
- [Background] Itzkovich M, Shefler H, Front L, Gur-Pollack R, Elkayam K, Bluvshtein V, Gelernter I, Catz A. SCIM III (Spinal Cord Independence Measure version III): reliability of assessment by interview and comparison with assessment by observation. Spinal Cord. 2018 Jan;56(1):46-51. doi: 10.1038/sc.2017.97. Epub 2017 Sep 12. PMID 28895576
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Mostafa, M. A., Plastow, A. N., and Savin-Baden, M. (2019). The effectiveness of spinal cord injury ADL inpatient education on rehabilitation outcomes: A systematic review and meta-analysis. British Journal of Occupational Therapy, 83,(1), 15-28. DOI: 10.1177/0308022619879019
- [Background] Mostafa, M. A., Plastow, A. N., and Savin-Baden, M. (2020). Developing of an Evidence-Informed Activities of Daily Living Educational Manual. Manuscript submitted for publication
- [Background] Polit, D. F., Beck, C. T. and Hungler, B. P. (2001). Essentials of Nursing Research: Methods, Appraisals, and Utilization. Fifth edition.: Lippincott, USA.
- [Background] Quittner, A. L., Espelage, D. L., Ievers-Landis, C., & Drotar, D. (2000). Measuring adherence to medical treatments in childhood chronic illness: Considering multiple methods and sources of information. Journal of Clinical Psychology in Medical Settings, 7(1), 41-54. https://doi.org/10.1023/A:1009545319673
- [Background] Wasson JH. Practice Standards for Effective Telemedicine in Chronic Care Management After COVID-19. J Ambul Care Manage. 2020 Oct/Dec;43(4):323-325. doi: 10.1097/JAC.0000000000000355. No abstract available. PMID 32858735
- [Result] Anderson K, Aito S, Atkins M, Biering-Sorensen F, Charlifue S, Curt A, Ditunno J, Glass C, Marino R, Marshall R, Mulcahey MJ, Post M, Savic G, Scivoletto G, Catz A; Functional Recovery Outcome Measures Work Group. Functional recovery measures for spinal cord injury: an evidence-based review for clinical practice and research. J Spinal Cord Med. 2008;31(2):133-44. doi: 10.1080/10790268.2008.11760704. PMID 18581660
- [Result] Chou HK, Lin IC, Woung LC, Tsai MT. An empirical study on outpatients' health education needs and the effectiveness of e-learning. Health Promot Pract. 2012 Jan;13(1):133-9. doi: 10.1177/1524839910385896. Epub 2010 Dec 29. PMID 21191081
- [Result] Letts L, Martin Ginis KA, Faulkner G, Colquhoun H, Levac D, Gorczynski P. Preferred methods and messengers for delivering physical activity information to people with spinal cord injury: a focus group study. Rehabil Psychol. 2011 May;56(2):128-37. doi: 10.1037/a0023624. PMID 21574732
- [Result] May L, Day R, Warren S. Evaluation of patient education in spinal cord injury rehabilitation: knowledge, problem-solving and perceived importance. Disabil Rehabil. 2006 Apr 15;28(7):405-13. doi: 10.1080/09638280500192439. PMID 16507503
- [Result] Scivoletto G, Tamburella F, Laurenza L, Molinari M. The spinal cord independence measure: how much change is clinically significant for spinal cord injury subjects. Disabil Rehabil. 2013 Oct;35(21):1808-13. doi: 10.3109/09638288.2012.756942. Epub 2013 Jan 24. PMID 23343359
- [Result] Shepherd JD, Badger-Brown KM, Legassic MS, Walia S, Wolfe DL. SCI-U: e-learning for patient education in spinal cord injury rehabilitation. J Spinal Cord Med. 2012 Sep;35(5):319-29. doi: 10.1179/2045772312Y.0000000044. PMID 23031169
- [Result] Wirth B, van Hedel HJ, Kometer B, Dietz V, Curt A. Changes in activity after a complete spinal cord injury as measured by the Spinal Cord Independence Measure II (SCIM II). Neurorehabil Neural Repair. 2008 May-Jun;22(3):279-87. PMID 18496904
- [Derived] Abu Mostafa M, Plastow NA, Savin-Baden M, Ayele B. The Impact of an Evidence-Informed Spinal Cord Injury Activities of Daily Living Education Manual (SADL-eM): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jul 22;11(7):e30611. doi: 10.2196/30611. PMID 35867399

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04735887/Prot_SAP_000.pdf